CLINICAL TRIAL: NCT05982691
Title: National Cancer Center Korea
Brief Title: Development of Asian Consortium for Data Collection and Clinical Trial of CNS Tumors
Status: Recruiting | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Joo-Young Kim, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC22-0194
Record Dates: First submitted 2023-05-30; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: CNS Germinoma; CNS Tumor; Asian Consortium
Keywords: CNS germinoma; CNS Tumor; Asian Consortium
MeSH Terms: conditions — Germinoma; Central Nervous System Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation Therapy(General guideline) Patients will receive radiotherapy after induction chemotherapy or right after diagnosis without diagnosis. The dose and fields of radiation will be according to the histology, presence of dissemination, and response to the induction chemotherapy or radiotherapy. Radiation therapy can be administered using either of photons or protons. When induction chemotherapy is administered, radiotherapy is recommended to be started within 6 weeks from the last chemotherapy.

SUMMARY:
<Purpose of the Research>

* Primary Establishing an Asian consortium to establish a database of pediatric CNS tumors in the prospective manner The target disease of this research focuses on pediatric tumors, and initially the registration of patients with CNS GCT will begin first.
* Secondary Developing clinical protocols for pediatric CNS tumors based in Asia

<Duration of Research Participation> Registration period for research subjects: 2022-08-01 - 2027-12-31 Duration of medical records to be utilized: to 2030-12-31 Total projected duration of research: IRB approved to 2032-12-31 Interim assessment of data quality and integrity: 6 Mo after Data collection Evaluation for the Adaptation of Protocols: 1 and 2 years after the initiation of the study Analysis of Quality of Life and other questionnaires: 3 and 5 years Interim Analysis of all data: 5 years (2027) Final analysis of treatment outcome: 2032

DETAILED DESCRIPTION:
<Selection standards>

* A patient who was diagnosed with CNS GCT and agreed to participate in the research between 2022-2027.

  * Patients diagnosed between 2016-2022 can be enrolled if the participating institute has IRB approval for recruiting these patients as separate IRB document (Seoul Asan Hospital) or by comprehensive IRB document (Singapore NCC, Taiwan Medical University), or by recruitment on the basis of acquirement of the consent form for research (NCC, Korea).

    * The age at the time of diagnosis is 0< ≤40 years

      * A patent who has been diagnosed with the relevant tumor via an operation or a biopsy ⑤In the case of CNS germinoma, a biopsy may not have been performed on a patient. In this case, the patient may register as germinoma if he or she meets the following criteria: -Germinoma is strongly suspected radiologically, and a tumor marker from serum or cerebrospinal fluid (CSF) has not increased above the institute's reference normal value;

        * Germinoma is suspected radiologically, and a tumor marker from serum or CSF has elevated above the institute's reference normal value (tumor markers may be AFP or hCG)

<Exclusion criteria> ①The patient or the guardian of the patient did not consent to participate.

<Attrition criteria>

* The patient refuses the treatment plan when the treatment is not completed.

  * The consent to participate has been rescinded in the process of data collection after the completion of the treatment.

    ③The research subject expresses the intention to rescind the consent to participate after the subject reaches the age of majority.

<Recruitment through an international multi-agency network> Managers at Korean institutions who agreed to participate in the research are charged with the registration of patient information. Internationally, researchers in each institution in Singapore, Taiwan, Thailand, and Korea which agreed to participate in the research enter the information by logging into a registration system.

Each institution obtained approval from its respective institutional review board.

ELIGIBILITY:
Inclusion Criteria:

* A patient who was diagnosed with CNS GCT and agreed to participate in the research between 2022-2027.

  * Patients diagnosed between 2016-2022 can be enrolled if the participating institute has IRB approval for recruiting these patients as separate IRB document (Seoul Asan Hospital) or by comprehensive IRB document (Singapore NCC, Taiwan Medical University), or by recruitment on the basis of acquirement of the consent form for research (NCC, Korea).

    * The age at the time of diagnosis is 0< ≤40 years

      * A patent who has been diagnosed with the relevant tumor via an operation or a biopsy ⑤ In the case of CNS germinoma, a biopsy may not have been performed on a patient. In this case, the patient may register as germinoma if he or she meets the following criteria: -Germinoma is strongly suspected radiologically, and a tumor marker from serum or cerebrospinal fluid (CSF) has not increased above the institute's reference normal value; -Germinoma is suspected radiologically, and a tumor marker from serum or CSF has elevated above the institute's reference normal value (tumor markers may be AFP or hCG)

Exclusion Criteria:

① The patient or the guardian of the patient did not consent to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Looking at the experience of collecting data for joint research in the Asian region, the number of patients data collected by all institutes including from Singapore, Taiwan, Korea and Japan during a 20-year period (1995-2015) were around 450 for germinoma, and 250 for mixed germinoma. Therefore, the projected collection of patient information from 10 institutes of 4 countries during the 5 years from 2022 to 2027 will be at a similar level, with around 400 patients, combined with two diseases.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic and diagnostic elements | Untill the year 2027
  * Sex, date of birth, birth order, weight at birth, education, disability diagnosis, parents' socio-economic information, cancer family history
  * Age at diagnosis, date of diagnosis, name of diagnosis, pathological name of the diagnosis, ECOG performance status at the time of diagnosis, location of tumor, stage, tumor marker, biopsy, etc.
Laboratory and pathologic assessments | Untill the year 2027
  * Laboratory assessments include full blood count, PT, PTT, serum electrolytes, alakaline phosphatase, alanine transferase, aspartate aminotransferase, bilirubin, serum creatinine, GFR, serum lactate, and ammonium.
  * Both of serum and CSF tumor markers including bHCG and AFP are highly recommended to be obtained at the time of diagnosis. Tumor markers in both serum and CSF should be obtained within 3 months after the completion of radiotherapy for final response evaluation.
  * Biopsy is strongly recommended as a component of diagnostic assessments, even when germinoma is highly suspected based on radiological images and tumor markers. Biopsy is particularly strongly recommended when ß-HCG is higher than 50 mIU/mL.
Radiological assessments | Untill the year 2027
  * Brain and spinal MRI with gadolinium contrast should be obtained at the time of diagnosis.
  * For early response evaluation, brain MRI is highly recommended to be obtained at radiation dose of 20 Gy in patients who are not given induction chemotherapy. Otherwise, brain MRI should be obtained after induction chemotherapy and before the initiation of radiotherapy.
  * For final response evaluation, brain MRI should be obtained within 3 months after the completion of radiotherapy.
Radiologic response criteria | Untill the year 2027
  * Complete response (CR): complete disappearance of visible disease on imaging. allowing for minimal residual disease/enhancement ≤0.5 cm maximal dimension in suprasellar or ≤1cm in pineal locations.
  * Partial response (PR): > 0.5 cm dimension residual in the suprasellar area or > 1 cm residual in pineal location, but ≥ 65% decrease in the sum of the products of the three perpendicular diameters (volume) of all target lesions.
  * Stable Disease (SD): Neither sufficient decrease in the sum of the products of the three perpendicular diameters of all target lesions to qualify for PR (taking as reference the initial baseline measurements), nor sufficient increase in a single target lesion to qualify for PD, and residual disease of > 1.5 cm maximal diameter.
  * Progressive Disease (PD): 40% or more increase in the product of perpendicular diameters (volume) of any target lesion, or the appearance of one or more new lesions.
Treatment elements | Untill the year 2027
  * Whether the operation has been performed and the extent of operation if performed
  * Chemotherapy: Medication used for treatment, treatment response, the timing of treatment (pre- or post-radiation therapy)
  * Radiation therapy: Site of treatment, treatment volume (radiotherapy field), radiation dose, treatment response, start date, end date
Treatment response, acute and late complications, and survival | Untill the year 2027
  * Treatment response (by radiologic imaging, tumor markers), treatment-related acute and late complications, co-morbid condition, last traced date, whether the patient survived or not
  * Whether the disease relapsed, the date of relapse, the location of relapse (brain or spine, out or inside of final boost field, out or inside of whole ventricular field)
  * Development of second malignant neoplasm (SMN)

SECONDARY OUTCOMES:
Neurocognitive assessment | Untill the year 2027
  • Neurocognitive functions of patients are highly recommended to be assessed before the initiation of treatment (either chemotherapy or radiotherapy) and at 1 years post-treatment, and every 1-2 years thereafter after the completion of all treatment.
Quality of life assessment | Untill the year 2027
  • Under the standard treatment, conduct a survey before initial treatment either chemotherapy or radiotherapy, 1 years post-treatment, and every 1-2 years thereafter after the completion of all treatment (Those who underwent chemotherapy before radiotherapy need to undergo first survey before chemotherapy and additionally a second survey before radiotherapy)
  1. Pediatric brain tumor (7-12 yrs old, 13-18 yrs old): PED FACT-BRS, Child, Adolescent / Parent
  2. Pediatric Quality of Life 4.0 Generic Core Scale(7-12 yrs old, 13-18 yrs old) : PedsQL, Child, Adolescent / Parent
  3. Quality of Life-Cancer survivors quesionnaire( ≥19 yrs old): QOL-CS-K, adult
  4. Children's depression inventory (7-18 yrs old) : CDI
  5. Self-Esteem Inventory (7-18 yrs old) : SEI

CONTACTS AND LOCATIONS:
Overall Officials: Joo-young Kim, M.D., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea